CLINICAL TRIAL: NCT05132751
Title: Effect of a Machine Learning Ventilator Decision System Versus Standard Controlled Ventilation on in Critical Care: a Randomized Trial
Brief Title: Machine Learning Ventilator Decision System VS. Standard Controlled Ventilation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hu Anmin (Other)
Responsible Party: Sponsor-Investigator, Hu Anmin, The Second Clinical Medical College of Jinan University, The Second Clinical Medical College of Jinan University
Organization: The Second Clinical Medical College of Jinan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LL-KY-2021396
Record Dates: First submitted 2021-10-07; First posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Mechanical Ventilation; Critically Ill Patients

STUDY DESIGN:
Intervention Model Description: ventilator decision system
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Machine Learning Ventilator Decision System Ventilation
  Interventions: Device: Machine Learning Ventilator Decision System
- Group B (Active Comparator): Standard Controlled Ventilation
  Interventions: Device: Machine Learning Ventilator Decision System

INTERVENTIONS:
Device: Machine Learning Ventilator Decision System — Artificial intelligence ventilator system for personalized mechanical ventilation

SUMMARY:
Ventilator-induced lung injury is associated with increased morbidity and mortality. Despite intense efforts in basic and clinical research, an individualized ventilation strategy for critically ill patients remains a major challenge. However, an individualized mechanical ventilation approach remains a challenging task: A multitude of factors, e.g., lab values, vitals, comorbidities, disease progression, and other clinical data must be taken into consideration when choosing a patient's specific optimal ventilation regime. The aim of this work was to evaluate the machine learning ventilator decision system, which is able to suggest a dynamically optimized mechanical ventilation regime for critically-ill patients. Compare with standard controlled ventilation, to test whether the clinical application of the machine learning ventilator decision system reduces mechanical ventilation time and mortality.

ELIGIBILITY:
Inclusion Criteria:

1. only the first ICU stay was eligible;
2. adults ≥ 18 years of age on ICU admission;
3. estimate mechanical ventilation time ≥24 hours;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Mechanical ventilation time | through study completion, an average of 5 days

SECONDARY OUTCOMES:
Length of ICU stay time | through study completion, an average of 1 week
Length of hospital stay | through study completion, an average of 2 weeks
In-hospital mortality | through study completion, an average of 2 weeks

IPD SHARING:
Plan to Share IPD: Undecided